CLINICAL TRIAL: NCT04181801
Title: Subtotal Cholecystectomy for Complicated Acute Cholecystitis: a Multicenter Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 052.GME.2019.D
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Subtotal Cholecystectomy; Complicated Acute Cholecystitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Subtotal cholecystectomy — a surgical procedure in which more than the top half of the gallbladder is removed

SUMMARY:
We believe that subtotal cholecystectomy is a safe alternative to total cholecystectomy when the complicated gallbladder is encountered, resulting in decreased or equivalent risk of bile duct injury, major vascular injury, postoperative hemorrhage, infectious complications, and mortality. Additionally, we hope to further elucidate the expected outcomes of the varying subtypes of subtotal cholecystectomy in order to determine the safest approach, assuring the lowest need for secondary intervention, recurrent biliary disease, or need for a completion cholecystectomy.

DETAILED DESCRIPTION:
The first reported subtotal cholecystectomy occurred in 1955. Additional case reports and studies have been carried out, further defining this terminology as a method of avoiding misidentification injuries of the biliary system or portal vasculature when critical view of safety cannot be safely achieved. Recent data supports the safety of this decision, showing equivalent morbidity rates to total cholecystectomy in a large metanalysis of 1,231 patients. Importantly, only 4 of the 30 included studies were prospective in nature, allowing definition variability and inconsistent reporting of outcomes. Additional reports showed variable data regarding effect on hospital LOS, need for secondary intervention (including endoscopic retrograde cholangiopancreatography (ERCP), percutaneous drainage bilioma, or completion cholecystectomy), infectious complications, biliary or major vascular injury, and mortality. Some studies suggest that while subtotal cholecystectomy is associated with a decreased rate of bile duct injury and a lower conversion to open operation, this comes at the cost of increasing bile leak and recurrent biliary complications. Furthermore, the relatively recent distinction between fenestrating and reconstituting subtypes of subtotal cholecystectomy remain ill-defined in many of these studies, and outcomes between the two modalities remain variable across the literature. There is an obvious need for a head-to-head, prospective comparison between these subtypes to determine the safety and efficacy of the chosen intervention. To determine the impact of these differing techniques for subtotal cholecystectomy (namely reconstituting and fenestrating subtypes) as indicated by Tokyo Criteria (Table 1), for the management of the difficult cholecystectomy on short-term and long-term patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Preoperative definitive diagnosis of acute cholecystitis (Tokyo guideline: Table 1)

Exclusion Criteria:

* Pregnant patients
* Prior history of subtotal cholecystectomy
* Percutaneous cholecystostomy tube in place
* Preoperative diagnosis other than acute cholecystitis
* Symptomatic cholelithiasis
* Gallstone pancreatitis
* Choledocholithiasis
* Malignant/benign tumor
* Others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible cholecystectomy cases from October 2019 to October 2020 at MDMC will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-operative complications and mortality | oct 2019 - sept 2021
  Incidence of post-operative complications and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michal Truitt, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided